CLINICAL TRIAL: NCT07381101
Title: Trazodone Dose and the Risk of Serious Adverse Events in Older Adults With Low Kidney Function: A Population-Based Cohort Study Research Protocol
Brief Title: Trazodone and the Risk of Serious Adverse Events
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 2026 0906 635 001; ICES #2026 0906 635 001 (Other: ICES, Ontario, Canada)
Record Dates: First submitted 2026-01-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease (CKD); Older Adults (65 Years and Older)
Keywords: Chronic Kidney Disease (CKD); Trazodone; Adverse events; Safety; Cohort study; Pharmacoepidemiology
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Trazodone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low dose (25-75 mg/day) Trazodone: Residents of Ontario, aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m² but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for trazodone (low dose 25-75 mg/day) with a day supply ≥ 5 days at an outpatient pharmacy under Ontario Drug Benefit (ODB) program from January 1, 2008, to March 01, 2025. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once. If the investigators conduct the study in Alberta, the accrual period for Alberta will be determined.
  Interventions: Drug: Trazodone HCl
- High dose (>75-150 mg/day) Trazodone: Residents of Ontario, aged 66 years or older with low kidney funciton (an eGFR <45 mL/min per 1.73 m² but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for trazodone (high dose >75-150 mg/day) at an outpatient pharmacy with a day supply ≥ 5 days under Ontario Drug Benefit (ODB) program from January 1, 2008, to March 31, 2025. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once. If the investigators conduct the study in Alberta, the accrual period for Alberta will be determined.
  Interventions: Drug: Trazodone HCl

INTERVENTIONS:
Drug: Trazodone HCl — The primary exposure of interest will be oral trazodone at a dose >75-150 mg/day.

SUMMARY:
This is a population-based retrospective, new-user, active comparator cohort study assessing whether initiating a new outpatient prescription of trazodone (>75-150 mg/day) compared to a lower dose (25-75 mg/day) is associated with an increased 30-day risk of serious adverse events among older adults with low kidney function (eGFR <45 mL/min/1.73 m²) who are not receiving dialysis and have no history of kidney transplantation.

The primary outcome is a 30-day composite of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality.

DETAILED DESCRIPTION:
*Summary*

Background:

Trazodone is a triazolopyridine antidepressant classified as a serotonin antagonist and reuptake inhibitor. It antagonizes serotonin 5-HT2A and 5-HT2C receptors, weakly inhibits serotonin reuptake, and also antagonizes α-1-adrenergic and histaminergic receptors. The U.S. Food and Drug Administration has approved trazodone for the treatment of major depressive disorder, and it is commonly prescribed off-label for insomnia, especially in older adults.

Trazodone is metabolized by the liver and excreted through the kidneys as an inactive metabolite. In patients with low kidney function, especially older adults, trazodone can accumulate and increase the risk of developing serious adverse events.

The most common measure to assess kidney function in routine clinical care is the estimated glomerular filtration rate (eGFR), expressed in lab reports as mL/min/1.73 m2. A normal eGFR is >90 mL/min/1.73 m2, and a value <45 mL/min/1.73 m2 is considered to be low.

Prescribing references, product monographs, and other standard sources do not provide daily dose recommendations for trazodone in patients with low kidney function. As a result, trazodone is often initiated at standard doses in this population. However, trazodone has not been studied well in patients with low kidney function.

The investigators aim to conduct a population-based cohort study among older adults with low kidney function in Ontario, comparing the risk of serious adverse events among those initiating a higher (>75-150 mg/day) dose versus a lower (25-75 mg/day) dose of trazodone in the outpatient setting.

Methods:

In this population-based retrospective cohort study, eligible participants will include older adults (≥66 years) with eGFR <45 mL/min/1.73 m² (not receiving dialysis or having a history of kidney transplantation) from Ontario who were dispensed a new outpatient prescription for oral trazodone (25-150 mg/day) with a day supply of ≥5 days. In Ontario, accrual will occur between January 1, 2008, and March 1, 2025. Based on the prescribed daily dose, individuals will be divided into two groups: low-dose (25-75 mg/day) and high-dose (>75-150 mg/day). Propensity score weighting will be used to ensure both groups are well-balanced on a comprehensive set of measured baseline characteristics.

The primary outcome will be a 30-day composite of all-cause hospitalization, emergency department visit, and mortality.

*Background* Trazodone is commonly used for the management of insomnia in older adults with low kidney function, at variable daily doses ranging from 25 to 150 mg/day. Trazodone-related serious adverse events reported in the single patient case reports include respiratory arrest, coma, arrhythmias, hypotension, delirium, and extrapyramidal symptoms. Overall, safety data for trazodone in patients with low kidney function is very limited, highlighting the need for a population-based drug safety study to evaluate its real-world safety profile in this population and inform better patient care.

Understanding the risks of initiating higher versus lower doses of trazodone in older adults with low kidney function can be used to guide safe prescribing and better outcomes in this population.

*Objectives* Is there a higher 30-day risk of a composite outcome of all-cause hospitalization, or all-cause emergency visit, or all-cause mortality among older adults with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who initiate a high dose (>75-150 mg/day) versus a low dose (25-75 mg/day) trazodone in the outpatient setting?

*Study design and setting* The investigators propose a population-based retrospective cohort study using linked administrative health data from Ontario. If the Ontario cohort is small to generate reliable estimates, the investigators will augment the study by performing an analysis using Alberta health administrative data.

Data will be sourced from ICES (ices.on.ca). It offers secure, encrypted individual-level data for Ontario residents, all with universal access to hospital and physician services under a government-funded, single-payer healthcare system. The use of data in this study is authorized under section 45 of Ontario's Personal Health Information Protection Act, which does not require review by a research ethics board. The information needed for analyzing the primary outcomes is available across specific databases within the ICES system: data on all-cause hospitalizations are available in the Canadian Institute for Health Information Discharge Abstract Database, emergency visits in the National Ambulatory Care Reporting System, and mortality in the Registered Persons Database.

If the investigators proceed with conducting the study in Alberta and combining the findings with Ontario, the Alberta data will be accessed through the Alberta Kidney Disease Network (AKDN), this dataset ends in ~ 2021.

The investigators are publicly registering the study protocol and documenting the study description, design, and statistical analysis prior to conducting outcome analyses. The results of this study will be reported adhering to RECORD reporting guidelines.

*Study Population* The investigators will include all older adults (≥66 years) with an eGFR <45 mL/min per 1.73 m2 (not receiving dialysis or having a history of kidney transplantation) who received a new outpatient prescription for oral trazodone with an initial dose between 25 and 150 mg/day and a day supply of ≥5 days. The dispensing date of the prescription will serve as the index date, and only the first eligible prescription will be included to ensure unique cohort entry, and each individual can enter the cohort only once.

*Baseline Characteristics* Health records, census files, hospital discharge records, laboratory data, and physician claims will provide baseline variables, including demographic characteristics (such as age, sex, rurality, neighborhood income quintile), comorbidities, and medication use. Baseline comorbidities and healthcare utilization will be assessed using 5-year and 1-year look-back periods from the index date. Baseline medication use will be assessed within 120 days prior to the index date.

*Outcomes* Participant observation time will be censored at the time of the first occurrence of the outcome of interest, death (if not the outcome of interest), or 30 days after the index date, whichever comes first.

The primary outcome is a 30-day composite outcome of all-cause hospitalization, all-cause emergency visit, and all-cause mortality.

Secondary outcomes will include Components of the primary composite outcome: 30-day all-cause hospitalization, all-cause emergency visit, all-cause hospitalization or emergency visit, and all-cause mortality, each examined separately.

30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with fragility fracture (hip, femur, humerus, wrist/forearm, pelvis, and spine), falls, hypotension or syncope.

30-day hospital encounter (hospital admission or emergency visit) composite of atrial fibrillation/flutter, ventricular arrhythmia/sudden cardiac death, and other arrhythmia (including pacemaker insertion, palpitations, tachycardia unspecified, atrioventricular block, supraventricular tachycardia, other conduction disorders, implantable cardiac defibrillator).

30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with delirium or encephalopathy (disorientation, transient alteration of awareness, and other unspecified symptoms and signs involving cognitive function) or hospital admission with receipt of an urgent computed tomography scan of the head.

*Statistical analysis plan* Categorical variables will be summarized as frequencies and proportions, while continuous variables will be summarized as means with standard deviations (SD) or medians with interquartile ranges (IQR), as appropriate.

Baseline characteristics will be compared between the high-dose (>75-150 mg/day) and the low-dose (25-75 mg/day) groups using standardized mean differences (SMDs), with an absolute SMD greater than 10% considered indicative of a meaningful imbalance.

Balancing comparator group: The investigators will use inverse probability of treatment weighting (IPTW) on the propensity score to balance baseline characteristics between the high-dose (>75-150 mg/day) and low-dose (25-75 mg/day) groups, including known predictors of trazodone use.

Propensity scores will be generated using a multivariable logistic regression model with all baseline characteristics.

Average treatment effect in the treated (ATT) weights will be used, where patients in the low-dose group will be assigned weights calculated as (propensity score / [1 - propensity score]) and patients in the high-dose group will receive a weight of 1. This method will produce a weighted pseudo-sample of patients in the referent group, i.e., low-dose trazodone with a similar distribution of measured baseline characteristics as the high-dose trazodone group. Baseline characteristics will be compared between groups using standardized differences in both unweighted and weighted samples.

Regression analysis: To evaluate the primary outcome composite measure of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality, the investigators will apply a modified Poisson regression analysis to estimate the risk ratio (95% CI) and binomial regression to estimate the risk difference (95% CI) using the weighted cohort, with the low-dose trazodone group as the referent.

Secondary analyses:

The investigators will conduct independent testing for all secondary outcomes without adjusting for multiple comparisons. Each test will be performed and reported independently. In line with best practices, the primary outcome will be presented with its P-value, and the investigators will report all secondary outcomes using point estimates with 95% confidence intervals.

Secondary analyses:

The investigators will conduct independent testing for all secondary outcomes without adjusting for multiple comparisons. Each test will be performed and reported independently. In line with best practices, the primary outcome will be presented with its P-value, and the investigators will report all secondary outcomes using point estimates with 95% confidence intervals.

Additional analyses: The investigators plan to conduct six additional analyses.

1. Effect measure modification (EMM):

   For EMM, the investigators will expand our cohort to all the eGFR levels and categorize them into three groups: eGFR ≥60, 45-<60, and <45 mL/min/1.73 m2. Baseline characteristics between high-dose (>75-150 mg/day) and low-dose (25-75 mg/day) trazodone groups will be assessed using standardized differences for all renal function categories combined and then within each of three eGFR categories (≥60, 45-<60, and <45 mL/min/1.73 m²).

   To further balance baseline characteristics between high-dose and low-dose traodone groups, the investigators will apply the IPTW method (described above), based on propensity scores for all the eGFR categories combined and within each of the three eGFR categories.

   EMM on the absolute scale for the primary composite outcome (30-day composite outcome of all-cause hospitalization, all-cause emergency visit, or all-cause mortality) will be examined across three baseline eGFR categories.

   EMM will be assessed on both the additive and multiplicative scales.

   For additive interaction, the investigators will use binomial regression with an identity link to estimate risk differences, including an interaction term between low-dose and high-dose trazodone groups and eGFR strata.

   For multiplicative interaction, the investigators will use modified Poisson regression analysis to estimate risk ratios, including an interaction term between low-dose and high-dose trazodone groups and eGFR strata.
2. Our interest in examining the safety of trazodone in older adults with low kidney function is derived from high-throughput computing analysis in which the investigators executed 700+ population-based, new-user cohort studies, each comparing 74 acute (30-day) outcomes across strata of kidney function (PMID: 38186562). In this analysis, trazodone was compared against non-users; the investigators found signs of harm, prompting us to undertake the current study. High-throughput analysis was run using Ontario data from January 1, 2008, to March 1, 2020. To confirm results, when there is no overlap, the investigators will run our analysis restricting the cohort after March 1, 2020.

   Examine whether the association between high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone and the primary outcome is different (modified) in 2 period categories (the period before the end date of the high-throughput computing, and the period after the end date of the high-throughput computing).

   The investigators will perform analysis restricted to the non-overlap period, i.e., after March 1, 2020.
3. Compute the hazard ratio for all outcomes within 30 days, illustrating the effect of the intervention on each outcome over time. The investigators expect hazard ratios results similar to risk ratios. Although the difference between hazard ratios and risk ratios may be minimal over a short follow-up period, the hazard ratio offers additional insight by accounting for time-to-event analysis.
4. Compare trazodone users (low-dose and high-dose separately) with non-users of trazodone to contextualize the magnitude and direction of risk observed in the dose-comparison analysis. This analysis will follow a new-user design and apply propensity score weighting to balance baseline characteristics between trazodone users and non-users.
5. The investigators will perform E-value analyses to determine the minimum association strength an unmeasured confounder would need with both the prescription drug and the outcome of interest (while adjusting for measured covariates) to eliminate the observed association.
6. Among patients with low kidney function (eGFR <45 mL/min/1.73 m²), the investigators will conduct prespecified subgroup analyses to examine whether the association between high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone and the primary 30-day composite outcome differs across clinically relevant subgroups. Subgroups will be defined by baseline eGFR category (<45-30 and <30 mL/min/1.73 m²), baseline opioid use, baseline benzodiazepine use, long-term care residence, depression, and dementia. Effect measure modification will be assessed on both the additive and multiplicative scales using interaction terms in weighted regression models.

*Combining Outcome Results from Ontario and Alberta* This approach will only be used if the investigators proceed with conducting the analysis in Alberta.Privacy-preserving methods:The investigators plan to use a privacy-preserving Cox-based approach for estimating risk ratios for multisite studies where individual-level data cannot be shared due to privacy constraints described by Shu et al. (2025). The proposed method requires only a single transfer of summary-level outputs from each province to the research team. It produces results identical to those from a corresponding log-binomial regression with combined individual-level data. The method was developed by adapting the risk-set table approach for survival outcomes, assuming stratified province-specific baseline risks, and allowing for confounding mitigation strategies such as propensity score matching or weighting to be done individually in each province. Each province will independently calculate these summary tables using its individual-level data. The summary-level risk-set tables generated in Alberta will be shared in a single data transfer to the coordinating site's analyst, where they will be used to estimate the combined risk ratios and 95% confidence intervals. This will enable a robust and consistent analysis while maintaining data privacy and adhering to regulatory compliance. To comply with privacy regulations for minimizing the chance of identification of any individual, in all manuscripts, numbers of individuals are suppressed in the case of 5 or fewer participants (reported as ≤5). All team members will sign any required data confidentiality and data use agreements.

ELIGIBILITY:
Inclusion Criteria:

The cohort will will include all older adults (≥66 years) with an eGFR <45 mL/min per 1.73 m2 (not receiving dialysis or having a history of kidney transplantation) who received a new outpatient prescription for oral trazodone with an initial dose between 25 and 150 mg/day and a day supply of ≥5 days between January 1, 2008 to March 1, 2025. The age criterion is set to guarantee that individuals in this population have had at least one year of prior prescription drug coverage. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once.

Exclusion Criteria:

1. Individuals with missing administrative database number, missing or invalid age (<0 or >105 years), missing or invalid sex, death on or before the index date, non-Ontario resident (for Ontario data), or non-Alberta residents (for Alberta data).
2. Individuals less than 66 years of age on the index date.
3. Those with evidence of any study drug prescription 180 days before the index date (to restrict to new users only).
4. Individuals with more than one study drug prescription on the index date, as this complicates the ability to ascertain the prescribed dose accurately.
5. Individuals with end-stage renal disease, chronic dialysis, or a kidney transplant prior to the index date.
6. Evidence with hospital discharge or emergency department visit in the two days prior to or on the index date to ensure a new outpatient prescription.
7. Individuals with no serum creatinine lab value in the 0-365 days prior to the index date.
8. Individuals with unstable baseline kidney function:

   If the most recent serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] <refer to this as test date 1>, and there is not at least one 'outpatient' serum creatinine in the year before test date 1, OR If the most recent prior serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] <refer to this as test date 1>, and while there is at least 'outpatient' serum creatinine test in the year before <test date 1>, the most recent outpatient test prior to <test date 1> differs by an eGFR 10 mL/min/1.73 m2 or more from the value on <test date 1>.

   In Ontario, it has been shown that outpatient serum creatinine measurements in the province, conducted on a single occasion, indicate stable values.
9. Individuals receiving palliative care in the 0-365 days prior to the index date, in this setting, dosing is less relevant; rather, the focus is comfort care.

The investigators restrict to the first prescription in individuals with more than one eligible prescription. Date of this prescription will be the index date (the Date from which the outcomes start being assessed).

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 66 years or older with low kidney function (eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new outpatient prescription for trazodone with a dose range of 25-150 mg/day and a day supply of ≥5 days between 2008 and 2025 in Ontario.
Sampling Method: Non-Probability Sample
Enrollment: 31459 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with a composite outcome of all-cause hospitalization or all-cause emergency visits, or all-cause mortality. | Older adults exposed to high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone will enter the cohort and be followed until the study outcome (first event), death, or 30 days from the cohort entry date.
  All-cause hospitalization, all-cause emergency visits, and all-cause mortality will be combined into a composite measure. Only the first hospitalization or first emergency department visit occurring within 30 days after the cohort entry date will be considered.

SECONDARY OUTCOMES:
Number of participants with all-cause hospitalization. | Older adults exposed to high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone will enter the cohort and be followed until the study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause hospitalization, individually presented as a secondary outcome. Only the first hospitalization after the cohort entry date will be considered.
Number of participants with all-cause emergency department visit. | Older adults exposed to high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone will enter the cohort and be followed until the study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause emergency department visit, individually presented as a secondary outcome. Only the first emergency department visit after the cohort entry date will be considered.
Number of participants with all-cause mortality | Older adults exposed to high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone will enter the cohort and be followed until the study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause mortality, individually presented as a secondary outcome.
30-day composite outcome of a hospital encounter with fragility fracture, falls, hypotension, or syncope. | Older adults exposed to high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone will enter the cohort and be followed until the study outcome (first event), death, or 30 days from the cohort entry date.
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with fragility fracture (hip, femur, humerus, wrist/forearm, pelvis, and spine), falls, hypotension, or syncope.
30-day composite outcome of a hospital encounter with delirium, encephalopathy, or hospital admission with receipt of an urgent computed tomography scan of the head | Older adults exposed to high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone will enter the cohort and be followed until the study outcome (first event), death, or 30 days from the cohort entry date.
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with delirium or encephalopathy (disorientation, transient alteration of awareness, other and unspecified symptoms and signs involving cognitive function) or hospital admission with receipt of an urgent computed tomography scan of the head.
30-day hospital encounter composite of atrial fibrillation/flutter, ventricular arrhythmia/sudden cardiac death, and other arrhythmia. | Older adults exposed to high-dose (>75-150 mg/day) versus low-dose (25-75 mg/day) trazodone will enter the cohort and be followed until the study outcome (first event), death, or 30 days from the cohort entry date.
  30-day hospital encounter (hospital admission or emergency visit) composite of atrial fibrillation/flutter, ventricular arrhythmia/sudden cardiac death, and other arrhythmia.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The dataset from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). The full dataset creation plan and underlying analytic code are available from the authors upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Background] Shu D, Zou G, Hou L, Petrone AB, Maro JC, Fireman BH, Toh S, Connolly JG. A simple Cox approach to estimating risk ratios without sharing individual-level data in multisite studies. Am J Epidemiol. 2025 Jan 8;194(1):226-232. doi: 10.1093/aje/kwae188. PMID 38973755
- [Background] Bathini L, Jeyakumar N, Sontrop J, McArthur E, Kang Y, Luo B, Bello A, Collister D, Ahmed S, Kaul P, Youngson E, Braam B, Melamed N, Hladunewich M, Garg AX. Impact of Baseline Kidney Function on the Rate of Progressive Kidney Disease After Pregnancy: A Population-Based Cohort Study Research Protocol. Can J Kidney Health Dis. 2025 Feb 28;12:20543581251318836. doi: 10.1177/20543581251318836. eCollection 2025. PMID 40027936
- [Background] Abdullah SS, Rostamzadeh N, Muanda FT, McArthur E, Weir MA, Sontrop JM, Kim RB, Kamran S, Garg AX. High-Throughput Computing to Automate Population-Based Studies to Detect the 30-Day Risk of Adverse Outcomes After New Outpatient Medication Use in Older Adults with Chronic Kidney Disease: A Clinical Research Protocol. Can J Kidney Health Dis. 2024 Jan 6;11:20543581231221891. doi: 10.1177/20543581231221891. eCollection 2024. PMID 38186562
- [Background] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648